CLINICAL TRIAL: NCT01981304
Title: Effects of a rapamycIn-eluting carboNized Stent With a Completely biodEgradable polymeR Coating on inflammaTory Biomarkers and Endothelial Damage
Brief Title: Effects of a rapamycIn-eluting carboNized Stent With a Completely biodEgradable polymeR Coating
Acronym: INERT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Other Study IDs: 807/2013/D
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DES with a biodegradable polymer coating: Patients receiving the first carbonized bio-absorbable coated rapamycin-eluting coronary stent at time of percutaneous coronary intervention

SUMMARY:
Percutaneous coronary intervention with stenting may induce endothelial damage/dysfunction and inflammatory reactions, which in turn delay healing and endothelialization and may lead to the occurrence of major adverse cardiac events (MACE), such as restenosis, atherosclerosis, and stent thrombosis.

Drugs, platforms and polymers are considered the protagonists of these pathophysiologic processes.

The objectives of the INERT study is to assess the extent of inflammation and endothelial damage induced by the first carbonized bio-absorbable coated rapamycin-eluting coronary stent at time of percutaneous coronary intervention and correlate the extent of these abnormalities with short and long-term clinical outcome and post-procedural evaluation of success.

As part of the study, a randomized sub-study will be carried out at the Coordinating Center in order to compare the biohumoral, clinical and procedural findings between patients with the carbonized bio-absorbable coated rapamycin-eluting coronary stent and those randomly assigned to receive stents with different platforms and polymers.

DETAILED DESCRIPTION:
Percutaneous coronary intervention with stenting may induce endothelial damage/dysfunction and inflammatory reactions, which in turn delay healing and endothelialization and may lead to the occurrence of major adverse cardiac events (MACE), such as restenosis, atherosclerosis, and stent thrombosis.

Drugs, platforms and polymers are considered the protagonists of these pathophysiologic processes.

Platforms Due to advances in stent technology, several stent platforms are now available, including the stainless steel, the cobalt-chromium, and the platinum-chromium stent series. Pre-clinical animal studies suggest that some platforms might have important advantages in terms of vascular compatibility and early and late healing. In a rabbit denudation model, it was shown that at 14 days the luminal surface area is incompletely endothelialised with the CrCo stents but nearly complete for other metals. Additionally, it has been shown that a thinner-strut stent is associated with reduced fibrin deposition and more rapid fibrin clearance in porcine coronary arteries compared with thicker stents, thus suggesting that the thin stent platforms may induce less injury. As a matter of fact, The second-generation DESs, with thinner struts, are obviously associated with a suppression of the neointimal response and a more rapid re-endothelialization but stainless steel based stent design might have a better conformability to the vessel wall which results to less malposition.

Polymers The polymer coating that elutes the antiproliferative drug has been linked to complications including delayed vessel healing, hypersensitivity reactions, atheroma, and restenosis, with the potential for repeat intervention, stent thrombosis, acute myocardial infarction, and sudden death.

The link between the permanent polymer and late adverse events has prompted the development of a variety of biodegradable polymer coatings. Absorption of the polymer may lower the rates of stent thrombosis, particularly beyond 1 year after stent implantation. In addition, stents with absorbable polymers may allow a shorter duration of dual antiplatelet therapy (DAPT) than currently recommended The incidence of late adverse events is likely to be lower after the absorption of the polymer than after the implantation of drug-eluting stents coated with a permanent polymer, as there is less ongoing inflammation than with permanent polymers. In a meta-analysis of randomized trials, metal stents that release an antiproliferative drug from an absorbable polymer coating had lower rates of MACE out to 4 years than metal stents that released a drug from a durable polymer. The randomized LEADERS (Limus Eluted from A Durable versus ERodable Stent) trial studies showed that a biolimus eluting stent coated with a biodegradable polymer had a lower risk of adverse cardiac events associated with very late ST through 5 years of follow-up, improving the long-term clinical outcomes compared with sirolimus-eluting stents coated with a durable polymer

Bio-absorbable coated Rapamycin-Eluting Coronary Carbonized Stent The new Rapamycin-Eluting Coronary Stent System is the first carbonized stent with a completely biodegradable polymer coating which contains rapamycin as drug for preventing early thrombotic and re-stenotic events. Absorption of carrier coating and drug takes place simultaneously within 6 weeks after implantation, leaving a carbonized stent platform behind. Because of the biodegradable polymer based technology, duration of the dual antiplatelet therapy after DES implantation might be shortened up to a few months.

The stent platform is a stainless stent that received CE-mark in 2001. It is a laser cut slotted tube, with multi-cellular design. The stent is characterized by a carbon-ion implanted layer (Inert Carbon Technology) that becomes incorporated within the metal lattice down to 0.05 mcm and avoids the leakage of heavy-metal ions as nickel and molybdenum. Usually, heavy metal ions released from stainless steel stent can cause allergic and inflammatory reactions which might be associated with in-stent restenosis. Conversely, the INERT-Technology alters common 316 stainless steel into a highly biocompatible alloy biodegradable polymer based sirolimus-eluting stent which is associated with earlier neointimal healing as compared to permanent polymer based eluting stent.

After carbonizing, the stent is coated with a thin layer of biodegradable polymer (PLGA). The coating is cleared from the stent in 45 to 60 days and and its degradation products (lactic and glycolic acid) are completely absorbed into the tissue within 90 days, leaving an inert bare metal stent, as confirmed during preclinical animal testing . This approach of drug delivery to the artery is aimed at achieving tissue coverage of the stent struts without excessive neointimal proliferation. Pre-clinical 'in vivo' studies have shown that the new Rapamycin-Eluting Coronary Stent System inhibit struts-associated inflammation and neointimal formation in the porcine coronary model.

Purpose

The objectives of the INERT study is to assess the extent of inflammation and endothelial damage induced by the first carbonized bio-absorbable coated rapamycin-eluting coronary stent at time of percutaneous coronary intervention and correlate the extent of these abnormalities with short and long-term clinical outcome and post-procedural evaluation of success.

As part of the study, a randomized sub-study will be carried out at the Coordinating Center in order to compare the biohumoral, clinical and procedural findings between patients with the carbonized bio-absorbable coated rapamycin-eluting coronary stent and those randomly assigned to receive stents with different platforms and polymers.

ELIGIBILITY:
Inclusion Criteria:

A de novo native coronary artery lesions (reference vessel diameter:2.5-3.75 mm) Class I indication to elective percutaneous coronary intervention Stable conditions and no recent acute coronary syndromes Normal baseline values of markers of myocardial damage (creatine kinase, creatine kinase-MB, myoglobin, and troponin I) Able to understand and willing to sign the informed CF

Exclusion Criteria:

Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary artery disease
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Post-PCI changes in markers of inflammation and endothelial damage | Baseline and 4 months after PCI
  Changes 4 months after PCI in indexes of endothelial damage (von Willebrand Factor, sE-selectin, Vascular cell adhesion molecule, Intercellular adhesion molecule) and inflammation (C-reactive protein, Fibrinogen, Plasminogen activator inhibitor, Interleukin-6)

SECONDARY OUTCOMES:
12-month rate of MACE | Up to 12 months
  12-months incidence of major adverse cardiac events (MACE-death, myocardial infarction, target vessel revascularization)

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Greco, MD, Study Chair — University Sapienza